CLINICAL TRIAL: NCT03627741
Title: A Pilot Study of Intralesional Injection of Triamcinolone Acetonide for Desmoid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Benjamin K. Wilke, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-008766
Record Dates: First submitted 2018-07-26; First posted 2018-08-13 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Fibromatosis
MeSH Terms: conditions — Fibroma | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Triamcinolone arm (Experimental): A concentration of 40 mg/ml of Triamcinolone Acetonide will be used for injections with a total dose of 120 mg of Triamcinolone given per injection. The injections will be performed under ultrasound guidance by a fellowship-trained musculoskeletal radiologist. The injection locations will be left to the discretion of the radiologist with the request to attempt to distribute the drug throughout the tumor. A total of three injections will be performed at six week intervals.
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Triamcinolone Acetonide — A concentration of 40 mg/ml of Triamcinolone Acetonide will be used for injections with a total dose of 120 mg of Triamcinolone given per injection. The injections will be performed under ultrasound guidance by a fellowship-trained musculoskeletal radiologist. The injection locations will be left to the discretion of the radiologist with the request to attempt to distribute the drug throughout the tumor. A total of three injections will be performed at six week intervals.

SUMMARY:
There is research supporting treatment of superficial fibromatoses (palmar fibromatosis and keloids) with triamcinolone acetonide injections. These lesions are histologically similar to deep fibromatoses (desmoid tumors). Currently there is little literature evaluating the response of desmoid tumors to injections of triamcinolone acetonide. The investigators aim to perform a pilot study evaluating the response of desmoid tumors to intralesional triamcinolone. If positive results are observed (based on RECIST criteria), then a phase II study will be initiated.

DETAILED DESCRIPTION:
Desmoid tumors are proliferations of fibroblasts and myofibroblasts, intermixed with abundant dense collagen. Histologically they are similar to superficial fibromatoses such as palmar (Dupuytren's disease) and plantar fibromatoses, as well as keloids. Unlike the superficial fibromatoses, desmoid tumors are located in the deep tissue and stratified based on an abdominal or extra-abdominal location.

There are currently many treatment options for desmoid tumors. Historically, wide surgical resection was the treatment of choice. This often resulted in a disfiguring appearance and recurrence was common, with rates between 30 - 40% following resection. Additionally, radiation and systemic therapies are performed, with an approximate 26% rate of objective response, based on RECIST. These therapies are however not without side effects. Observation initially is also a reasonable approach as a recent study reported up to 60% of desmoids demonstrating stable disease and 18% spontaneously regressing over a five year period. Longer follow-up studies are needed to determine the true natural history of desmoid tumors, but there currently is a need for an alternative treatment strategy with increased efficacy and fewer side-effects once observation has failed.

Corticosteroids, such as triamcinolone acetonide, have long been used in the treatment of hypertrophic scars and keloids in order to decrease the size of the lesion. Proposed mechanisms of action of corticosteroids on keloids and hypertrophic scars include a decrease in the production of collagen, dissolution of insoluble collagen (collagenolysis), a decrease in the local inflammatory process, and an increased rate of apoptosis of fibroblast and inflammatory cells. Recently, reports have evaluated the use of triamcinolone acetonide in Dupuytren's disease, a superficial fibromatosis. A randomized controlled trial evaluated range of motion in patients following needle aponeurotomy alone and in combination with serial triamcinolone injections. They found improved range of motion in the triamcinolone cohort up to 24 months following treatment. Similarly, Ketchum et al reported that 97% of Dupuytren's nodules showed clinical regression following an average of 3.2 intralesional injections with triamcinolone acetonide, although half of these patients did experience reactivation of the disease at 1-3 years following treatment.

Currently there is limited reported experience with treatment of desmoid tumors by steroid therapy. Rhee et al reported a case of a chest wall desmoid tumor that recurred after two surgical resections and postoperative radiation therapy. They treated the lesion with weekly intralesional injections of 120 mg of triamcinolone acetonide for 4 weeks. At six months they noted a reduction in the size of the lesion. Similarly, Umemoto et al. reported a case of a 37 year old male with familial polyposis coli and intra-abdominal desmoid tumors. He was treated with oral prednisolone therapy with gradual regression of the lesions. At one year and six months following his last operation, the patient had no signs of recurrence of the desmoid tumors.

Based on this background information we aim to perform a pilot study of 10 patients with a histologically confirmed diagnosis of extra-abdominal aggressive fibromatosis (desmoid tumor) in order to determine the response rate of intralesional injections of triamcinolone acetonide. Response will be evaluated using the World Health Organization (WHO) response criteria, total volume of the tumor, T2 signal hyperintensity, and RECIST.

ELIGIBILITY:
Inclusion Criteria

1. Patients with histologically confirmed diagnosis of extra-abdominal aggressive fibromatosis (desmoid tumor).
2. At least one of the following: Desmoid tumor that has shown stability in size over consecutive axial imaging (CT or MRI) at least 3 months apart AND presence of any tumor-related symptoms OR an increase in size based on consecutive axial imaging (CT or MRI). Additionally, for patients with a desmoid tumor which has been irradiated, at least a 10% increase in size by volume since receiving radiotherapy is required.
3. ECOG Performance status of < 1.
4. Able to participate in three guided injection procedures.
5. Able to undergo a MRI with and without contrast of the tumor site.
6. Age > 18 years and ≤ 89 years.
7. Willing to sign an informed consent form.
8. Willing to comply with protocol procedures including required 21 month follow up after last injection.

Exclusion Criteria

1. Allergy to the test drug or a component of its formulation
2. Patients with a desmoid tumor which has been stable in size and without symptoms or decreased in size over the prior three months utilizing axial imaging according to the following criteria; (a) 10% when comparing a prior CT scan to a current MRI, or (b) more than 5% when comparing a prior MRI to a current MRI.
3. The patient must not be on anticoagulation (Aspirin okay)
4. The patient should not be pregnant or trying to become pregnant, and willing to use adequate contraception during study participation to avoid pregnancy
5. The patient should not be breastfeeding
6. Active infection that in the opinion of the investigator compromises the patient's participation (i.e., a UTI is ok)
7. A diagnosis of idiopathic thrombocytopenia purpura
8. Undergoing concomitant treatment (including radiation, systemic treatment, surgery, or other tumor directed therapy). The patient must be off of the systemic therapy for a period of at least 5 drug half-lives prior to enrolling in the study.
9. Uncontrolled or poorly controlled diabetes mellitus
10. Has an uncontrolled illness including, but not limited to, uncontrolled infection, or psychiatric illness/social situations that in the opinion of the investigator would limit compliance with study requirements

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Response rate of desmoid tumors to serial triamcinolone injections based on WHO criteria. | 2 years
  Based on MRI imaging
Response rate of desmoid tumors to serial triamcinolone injections based on change in tumor volume. | 2 years
  Based on MRI imaging
Response rate of desmoid tumors to serial triamcinolone injections based on change in T2 signaling hyperintensity. | 2 years
  Based on MRI imaging
Response rate of desmoid tumors to serial triamcinolone injections based on RECIST. | 2 years
  Based on MRI imaging

SECONDARY OUTCOMES:
Number patients experiencing a non-serious adverse event following triamcinolone injections. | 6 months following initial administration of triamcinolone injections
  Defined as any untoward or undesirable experience associated with the use of a medical product.
Number of patients experiencing a serious adverse event following triamcinolone injections. | 6 months following initial adminstration of triamcinolone injections.
  Including hospitalization, prolonged disability/incapacity, life-threatening adverse experience, birth defect, and death.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin K Wilke, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials